CLINICAL TRIAL: NCT07125170
Title: Immersive Virtual Reality in Cognitive Rehabilitation of Patients With Post-Stroke Cognitive Impairment: A Pilot Study at the Department of Physical Medicine and Rehabilitation, Clinical Hospital of the University of Chile
Brief Title: Immersive Virtual Reality in Cognitive Rehabilitation of Patients With Post-Stroke Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Natalia Gattini, Asistant professor, University of Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1497/25
Record Dates: First submitted 2025-07-29; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Post-Stroke Cognitive Impairment (PSCI); Cognitive Dysfunction; Virtual Reality Therapy; Virtual Reality Cognitive Training; Cognitive Rehabilitation
Keywords: virtual reality; Cognitive rehabilitation; Immersive Therapy; Meta Quest 3; Kinesix XR; Occupational Therapy; Montreal Cognitive Assessment (MoCA); Simulator Sickness Questionnaire (SSQ)
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a pilot, prospective, interventional, uncontrolled clinical study with a single assigned group. All participants will receive immersive virtual reality cognitive rehabilitation (Meta Quest 3, Kinesix XR application) for 30 minutes at the start of each occupational therapy session, followed by 30 minutes of conventional cognitive rehabilitation. Each participant will complete 10 sessions over an approximate period of 4 to 5 weeks. The study model is designed to assess the feasibility, safety, usability, and satisfaction of using immersive virtual reality in patients with post-stroke cognitive impairment, as well as its preliminary impact on cognitive function and quality of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-based Cognitive Rehabilitation (Experimental): Participants receive cognitive rehabilitation supported by immersive virtual reality using the Meta Quest 3 headset and the Kinesix XR application. Each session lasts 60 minutes, with the first 30 minutes involving VR-based cognitive tasks supervised by an occupational therapist. A total of ten sessions are completed over a period of approximately four weeks, with a frequency of two to three sessions per week. This arm is designed to assess the feasibility, safety, usability, and preliminary effects of VR-assisted rehabilitation in patients with post-stroke cognitive impairment.
  Interventions: Device: Kinesix XR on Meta Quest 3

INTERVENTIONS:
Device: Kinesix XR on Meta Quest 3 — Participants receive cognitive rehabilitation using immersive virtual reality through the Meta Quest 3 headset and the Kinesix XR application. Each session lasts one hour, with the first 30 minutes involving VR-based tasks guided by an occupational therapist. The intervention consists of a total of ten sessions, delivered two to three times per week. The VR component is integrated into the standard outpatient cognitive rehabilitation program. The study aims to evaluate the feasibility, safety, and acceptability of using this device during therapy.

SUMMARY:
This pilot study aims to evaluate the feasibility of implementing immersive virtual reality (VR) in cognitive rehabilitation for adults with post-stroke cognitive impairment receiving outpatient therapy. Participants will use a head-mounted display and interactive software to engage in gamified cognitive exercises that simulate memory, attention, and executive function tasks. The intervention consists of 10 sessions, delivered two to three times per week over a period of approximately four weeks. The study will assess multiple feasibility indicators, including the recruitment rate based on eligibility criteria, the safety and tolerability of VR sessions for participants, and the usability and satisfaction reported by occupational therapists administering the intervention. Additionally, exploratory outcomes include changes in global cognition and specific cognitive domains, as well as self-reported quality of life. Adverse effects related to VR use will be tracked. This pilot study will help inform the design and implementation of future, larger-scale clinical trials.

DETAILED DESCRIPTION:
This is a single-arm pilot study designed to evaluate the feasibility of implementing immersive virtual reality (VR) in cognitive rehabilitation for adults with post-stroke cognitive impairment. The study is conducted at the Occupational Therapy Unit of the Hospital Clínico Universidad de Chile and targets adult patients with documented cognitive impairment following a cerebrovascular accident (CVA).

Participants will undergo ten individual VR-assisted cognitive rehabilitation sessions, scheduled at a frequency of two to three sessions per week. Each session lasts approximately one hour, with the first 30 minutes incorporating immersive VR using the Meta Quest 3 headset and the Hand Physics Lab application. This application provides interactive cognitive exercises in a motivating and safe virtual environment. All sessions are supervised by occupational therapists trained in VR therapy.

The study aims to collect feasibility data, including recruitment rates based on inclusion and exclusion criteria, participant adherence to the intervention schedule, and reasons for withdrawal if any. Safety and tolerability will be assessed through patient-reported adverse effects (e.g., dizziness, nausea, or eye strain) using the Simulator Sickness Questionnaire (SSQ). Usability and satisfaction with the VR system will be evaluated from the perspective of the occupational therapists delivering the intervention.

Exploratory outcomes include changes in cognitive function measured with the Montreal Cognitive Assessment (MoCA) and in quality of life using the NeuroQoL short form. These measurements are taken before and after the intervention period. No compensation is provided for participation, and patients continue receiving standard care.

This pilot study does not aim to establish efficacy. Instead, it will provide essential data regarding the feasibility, safety, user experience, and preliminary clinical trends necessary to inform the development of future, larger-scale trials

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with a cerebrovascular accident of any etiology with less than 3 months of progression
* Patients with mild to moderate cognitive impairment post-stroke (impairment in at least one cognitive domain)
* MoCA score of less than 24 points
* Referred for cognitive rehabilitation at the Occupational Therapy Unit of HCUCH

Exclusion Criteria:

* Patients with refractive errors that prevent the use of the headset
* Patients with any type of aphasia that prevents the administration of the MoCA test
* Patients with severe psychiatric disorders (presence of psychotic symptoms or derealization)
* Patients with severe motor impairments (lack of trunk control or global strength of both upper limbs < M3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who complete ≥80% of planned sessions. | From first session to week 5 (after completion of the 10-session VR program)
  Number of participants who complete at least 8 of 10 sessions divided by total enrolled participants.
Incidence of VR-related adverse events requiring session interruption | From first session to week 5 (after completion of the 10-session VR program)
  Percentage of participants with one or more adverse events related to virtual reality that result in stopping a session, as documented in the patient's clinical record by the occupational therapist. Adverse events include, but are not limited to, nausea, dizziness, headache, and visual fatigue. In addition, symptoms associated with virtual reality will be monitored using the full Spanish-validated version of the Simulator Sickness Questionnaire (SSQ) after sessions 1, 5, and 10. The outcome measure will consider both sources of information -therapist-recorded clinical notes and SSQ scores- to identify and classify safety-related events.
Therapist-reported usability and satisfaction with immersive virtual reality in cognitive rehabilitation | At week 5 (after completion of the 10-session VR program)
  Therapist-reported usability and satisfaction with the immersive virtual reality intervention, measured using a custom-designed questionnaire rated on a 5-point Likert scale (1 = strongly disagree / very dissatisfied, 5 = strongly agree / very satisfied). The questionnaire includes five statements assessing ease of device setup, ability to personalize VR activities to the patient's cognitive needs, patient motivation during VR sessions, facilitation of active participation through immersion, and overall recommendation of the technology for cognitive rehabilitation. Total scores range from 5 to 25, with higher scores indicating greater usability and satisfaction. The questionnaire will be administered once, at week 5 (after completition of the 10-session VR program)

SECONDARY OUTCOMES:
Change in "Montreal Cognitive Assessment (MoCA)" score | Measured at baseline (before the intervention) and at week 5 (after completion of the 10-session VR program)
  Change in the "Montreal Cognitive Assessment (MoCA)" score (range 0-30, higher values indicate better cognitive function). The MoCA is a validated cognitive screening tool designed to detect mild cognitive impairment and assess multiple domains, including visuospatial/executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation. The Chilean validated version will be administered by a certified occupational therapist at two time points: at baseline (prior to the start of the intervention) and at week 5 (the end of the intervention period). The change will be calculated as the post-intervention score minus the baseline score.
Change in quality of life measured by NeuroQoL (Cognitive Function Short Form) | Measured at baseline (before the intervention) and at week 5 (after completion of the 10-session VR program)
  Change in the "Quality of Life in Neurological Disorders (Neuro-QoL) Cognitive Function Short Form" score (range 8-40, higher scores indicate better self-reported cognitive function and quality of life). The Cognitive Function Short Form is a validated patient-reported outcome measure designed to assess perceived cognitive abilities in adults with neurological conditions. For this study, the validated spanish version will be used. Participants will self-complete the questionnaire at two time points: at baseline (prior to starting the intervention) and at week 5 (after completing the 10-session immersive virtual reality cognitive rehabilitation program). The change will be calculated as the post-intervention score minus the baseline score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico de la Universidad de Chile, Independencia, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Pallesen H, Andersen MB, Hansen GM, Lundquist CB, Brunner I. Patients' and Health Professionals' Experiences of Using Virtual Reality Technology for Upper Limb Training after Stroke: A Qualitative Substudy. Rehabil Res Pract. 2018 Feb 8;2018:4318678. doi: 10.1155/2018/4318678. eCollection 2018. PMID 29593910
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699